CLINICAL TRIAL: NCT00756496
Title: A Multi-center Feature Analysis Study to Compare the Diagnostic Accuracy of Siemens' Image Processing (SIP) Algorithms With Lorad's Image Processing (LIP) Algorithms in Detecting and Characterizing Breast Lesions
Brief Title: Case Collection Study to Support Digital Mammography Image Software Change
Acronym: LIP2SIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Medical Solutions USA - CSG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SMS-SP04-06
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Mammography screening and diagnosis

INTERVENTIONS:
Device: Mammography screening and diagnosis — Mammography screening and diagnosis

SUMMARY:
The primary objective of this study is to compare image processing software to support a new image processing software application for a full-field digital mammography (FFDM) system.

ELIGIBILITY:
Inclusion Criteria:

* Female
* > 40 years

Exclusion Criteria:

* Pregnant women, or women who may become pregnant
* Mammographic evidence of breast surgery, prior radiation to the breast, needle projection or pre-biopsy markings are evident in the mammogram (but may include breast implants)
* Palpable lesion or one that is visible by another modality
* Inmates

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond C Duhamel, Ph.D., Study Director — Siemens Medical Solutions USA, Inc

RESULTS

PARTICIPANT FLOW:
Groups:
- Mammography Exam: Full Field Digital Mammography exam
Period: Overall Study
Arm/Group | Mammography Exam
Started | 442
Completed | 442
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FFDM Mammography Examination: Screening or diagnostic mammography exam.
Arm/Group | FFDM Mammography Examination
Number analyzed (Participants) | 442
Age, Customized [Count of Participants; unit: Participants]
  >=40 years old | 442
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 442
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 442

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Characteristic (ROC) Curve to Compare Diagnostic Accuracy of 2 Algorithms in Breast Cancer Diagnosis
Description: The primary objective of this study was to demonstrate non-inferiority of the Siemens' processing algorithm to Lorad's processing algorithm with regards to readers' diagnostic accuracy in detecting and characterizing breast lesions. The non-inferiority analyses were performed by comparing the area under the ROC curve (AUC) for the two algorithms & to compare false positive marks per subject.
  The ROC curve incorporates both sensitivity (true positive rate) and specificity (true negative rate) providing a single assessment incorporating both measures. It shows in a graphical way the trade-off between clinical sensitivity and specificity for every possible cut-off for a test, and gives an idea about the benefit of using the test in question. The higher the total area under the curve, the greater the predictive power of the reader assessments.
  A breast-based analysis was used for the primary AUC comparison in order to obtain additional power by having more normal/benign breasts.
Time Frame: ~1 year. Women with negative or biopsy benign findings at baseline (study entry) were followed for 1 year to confirm the negative status at 1-year follow-up mammography exam. Women diagnosed with cancer were not followed up.
Measure: Mean (Standard Error); unit: probability
Units Other Than Participants: breasts
Groups:
- FFDM Mammography Exam - LIP Algorithm: Screening or diagnostic Full Field Digital Mammography (FFDM) exam
- FFDM Mammography Exam - SIP Algorithm: The same 130 raw data images were externally reprocessed with the Siemens processing algorithm.
Arm/Group | FFDM Mammography Exam - LIP Algorithm | FFDM Mammography Exam - SIP Algorithm
Number analyzed (Participants) | 130 | 130
Number analyzed (breasts) | 260 | 260
probability | 0.884 (0.008) | 0.880 (0.008)

ADVERSE EVENTS:
Groups:
- Mammography Exam: FFDM screening or diagnostic mammography exam
Arm/Group | Mammography Exam
Serious Adverse Events (participants affected / at risk) | 0/442
Other Adverse Events (participants affected / at risk) | 0/442

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No